CLINICAL TRIAL: NCT02056067
Title: Hormones and Physical Exercise (HOPE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0906005263; CA132931 (Other: Other Federal ID)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Arthralgia
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): The exercise intervention group will receive social, behavioral support and research staff contact time to encourage them to increase their activity level to include twice weekly strength-training sessions and 150 min of walking/week (e.g., three 50-min walking sessions or five 30-min walking sessions) over 12 months.
  Interventions: Behavioral: Exercise
- Attention Control (Health Education) (Active Comparator): The Attention Control Group will be provided written information that emphasizes the importance of a healthy lifestyle. Participants will be encouraged to follow the NCI and ACS physical activity guidelines. This procedure was followed in our exercise trials, with no increase in physical activity levels observed at follow-up among women in the usual care group. Attention Control participants will also receive frequent contacts throughout the 12 month intervention. Each month, women randomized to attention control will be contacted by phone to discuss a health education topic of interest
  Interventions: Behavioral: Attention Control (Health Education)

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention group will receive social, behavioral support and research staff contact time to encourage them to increase their activity level to include twice weekly strength-training sessions and 150 min of walking/week (e.g., three 50-min walking sessions or five 30-min walking sessions) over 12 months.
  Arms: Exercise
Behavioral: Attention Control (Health Education) — The Attention Control Group will be provided written information that emphasizes the importance of a healthy lifestyle. Participants will be encouraged to follow the NCI and ACS physical activity guidelines. This procedure was followed in our exercise trials, with no increase in physical activity levels observed at follow-up among women in the usual care group. Attention Control participants will also receive frequent contacts throughout the 12 month intervention. Each month, women randomized to attention control will be contacted by phone to discuss a health education topic of interest
  Arms: Attention Control (Health Education)

SUMMARY:
The investigators propose to examine 121 postmenopausal women diagnosed with hormone-receptor positive breast cancer who have been taking aromatase inhibitors (AI) for at least 6 months and are experiencing at least mild arthralgia originating during AI treatment, the yearlong effect of exercise vs. attention control (health education), and on toxic side effects of AI.

DETAILED DESCRIPTION:
The investigators propose to examine, in 121 postmenopausal breast cancer survivors who have been taking an AI for at least 2 months and are currently experiencing at least mild arthralgia associated with AI use, the effect of a randomized controlled exercise intervention vs. attention control (health education) on severity of arthralgia, endocrine-related Quality of Life(QOL), Bone Mineral Density(BMD), and mediators/mechanisms influencing the effect of exercise on arthralgia severity. Women will be randomized to a year long exercise program or attention control group. Women randomized to exercise will participate in 150 min/wk of aerobic exercise and a twice-weekly strength training program. The investigators will conduct baseline, six-, and 12-month clinic visits, as well as a 3- and 9-month mailing to evaluate the effect of the intervention on study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (defined as the surgical or natural absence of menstrual cycles for at least 1 year prior to breast cancer diagnosis).
* 75 years or younger
* AJCC Stages I-IIIC Breast Cancer
* Taking an AI for at least 2 months
* Currently experiencing at least mild arthralgia (= or > 3 on the BPI) associated with AI use
* Physically able to exercise and physician consent to start an exercise program
* Sedentary activity pattern (< 90 mins/week of moderate-to-vigorous intensity sports activity) within the past year and low fitness level
* No more than one strength training session per week within the past year
* Agrees to be randomly assigned to either exercise or attention control
* Gives informed consent to participate in all study activities
* Able to come for baseline, 6-, and 12-month clinic visits and strength training sessions (6-month intervention study - able to come for baseline, 6-month clinic visits and strength training sessions).
* Mentally competent

Exclusion Criteria:

* Lymphedema with self reported 'flare up' in the past 4 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Arthralgia Severity | 6 months
  Measured using the Brief Pain Inventory (BPI). Subjects are asked to rate pain by circling a number from 0-10 that describes pain at its "worst", "least", and "average" with 0 being no pain and 10 being "pain as bad as you can imagine".
Change from Baseline in Arthralgia Severity | 12 months
  Measured using the Brief Pain Inventory (BPI). Subjects are asked to rate pain by circling a number from 0-10 that describes pain at its "worst", "least", and "average" with 0 being no pain and 10 being "pain as bad as you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Irwin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Thomas GA, Cartmel B, Harrigan M, Fiellin M, Capozza S, Zhou Y, Ercolano E, Gross CP, Hershman D, Ligibel J, Schmitz K, Li FY, Sanft T, Irwin ML. The effect of exercise on body composition and bone mineral density in breast cancer survivors taking aromatase inhibitors. Obesity (Silver Spring). 2017 Feb;25(2):346-351. doi: 10.1002/oby.21729. Epub 2016 Dec 27. PMID 28026901
- [Derived] Irwin ML, Cartmel B, Gross CP, Ercolano E, Li F, Yao X, Fiellin M, Capozza S, Rothbard M, Zhou Y, Harrigan M, Sanft T, Schmitz K, Neogi T, Hershman D, Ligibel J. Randomized exercise trial of aromatase inhibitor-induced arthralgia in breast cancer survivors. J Clin Oncol. 2015 Apr 1;33(10):1104-11. doi: 10.1200/JCO.2014.57.1547. Epub 2014 Dec 1. PMID 25452437